CLINICAL TRIAL: NCT04063683
Title: Paclitaxel and DDP Combined With Anlotinib in the First-line Treatment for Patients With Advanced Esophageal Squamous Cell Carcinoma: a Single Arm, Multicentre Trial.
Brief Title: Paclitaxel and DDP Combined With Anlotinib in the First-line Treatment for Patients With Advanced Esophageal Squamous Cell Carcinoma（ESCC）.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019315
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib with chemotherapy (Experimental)
  Interventions: Drug: Anlotinib Hydrochloride, Paclitaxel, cisplatin

INTERVENTIONS:
Drug: Anlotinib Hydrochloride, Paclitaxel, cisplatin — * anlotinib: 1 capsule (10mg) once a day, d1-d14 per cycle, 3 weeks for a treatment cycle.
  * Paclitaxel: intravenously infused at 135mg/ m2, administered d1 per cycle, 3 weeks for a treatment cycle.
  * Cisplatin: administered after paclitaxel, intravenously infused at 60-75 mg/m2, divided into d1-d3 medications per cycle; 3 weeks for one treatment cycle.

SUMMARY:
To evaluate the efficacy and safety of paclitaxel and DDP combined with Anlotinib in the treatment of advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* histopathology confirmed unresectable, locally recurrent or metastatic advanced esophageal squamous cell carcinoma (excluding mixed type adenosquamous carcinoma );
* Those who have not received systemic treatment before, or who relapsed after (new) adjuvant therapy/radical surgery more than 6 months ; Note: Including advanced or recurrent Patients who ever received only radiotherapy on non-target lesions. The duration from the end of palliative treatment for local lesions (non-target lesions) to enrollment should > 2 weeks;
* According to RECIST 1.1, at least one measurable lesion; the measurable lesions should not have received local treatment such as radiotherapy (for the lesions in the area where received local radiotherapy, it can also be regarded as a target lesion if confirmed to progress according to the recist1.1);
* Age from 18-75 years old;
* ECOG PS score: 0-1; expected survival time more than 3 months;
* Main organs function is normal;
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 3 months after study is stopped；the result of serum or urine pregnancy test should be negative before enrollment；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 2 months after study is stopped.
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Patients tends to have complete obstruction or patients requiring interventional treatment for obstruction;
* ulcerated esophageal squamous cell carcinoma patients;
* after esophageal or endotracheal stent implantation;
* Patients with a high risk of bleeding or perforation due to the apparent invasion of adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed fistulas;
* patients with ESCC who have not undergone surgical resection but have not reduced esophageal lesions after radiotherapy;
* allergic to paclitaxel and cisplatin preparations or excipients;
* Adjuvant chemotherapy patients who have used paclitaxel or cisplatin, and relapse or metastasize within one year;
* A variety of factors affecting oral medications (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
* The of liver metastases accounts for more than 50% of the total liver volume;
* patients with any severe and / or uncontrolled disease, including:Unsatisfactory blood pressure control using antihypertensive drugs (systolic blood pressure ≥150 mmhg or diastolic blood pressure ≥100) Mmhg) patients; patients with grade ≥ myocardial ischemia or myocardial infarction, arrhythmia (including qt interval ≥ 480ms); according to nyha criteria, iii-iv cardiac dysfunction, or cardiac ultrasonography prompted left ventricular ejection fraction (lvef) <50% of patients;live Severe infection that is sexual or uncontrolled;Liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis;poor diabetes control (fasting blood glucose (fbg)>10mmol/l);Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation > 1.0 g;
* long-term unhealed wounds or fractures;
* Patients with active hemorrhage within 2 months of primary lesions; pulmonary hemorrhage with NCI CTC AE grade >1, 4 weeks before of enrollment; other sites of bleeding NCI CTC AE grade >2, 4 weeks before of enrollment; patients with bleeding tendency (such as active gastrointestinal ulcers) or patients undergoing thrombolytic or anticoagulant therapy such as warfarin, heparin or its analogues;
* Have undergone major surgery (craniotomy, thoracotomy or open surgery) within 4 weeks prior to the first dose study or Major surgery is required during the study period.
* A history of gastrointestinal perforation and/or fistula occurred within 6 months prior to treatment; or an overactive/venous thrombosis event such as a cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and lung Embolism.
* Symptomatic central nervous system metastasis and/or cancerous meningitis are known to exist;
* Clinically significant ascites, including any ascites that can be found on a physical examination, ascites that has been treated or currently in need of treatment, and only those with a small amount of ascites but no symptoms can be selected;
* A moderate amount of fluid in both sides of the chest, or a large amount of fluid in one side of the chest, or has caused respiratory dysfunction Patient to be drained;
* known to have active tuberculosis;
* suffering from interstitial lung disease requiring steroid therapy;
* Uncontrolled metabolic disorders or other non-malignant tumors or systemic diseases or cancer secondary reactions that can lead to higher medical risks and/or survival Evaluation of uncertainty;
* Significantly malnourished patients;
* those who have a history of psychotropic substance abuse and are unable to quit or have a mental disorder;
* A history of immunodeficiency, including a positive HIV test or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
* History of other primary malignancies, but the following : 1) complete remission of malignant tumors for at least 2 years prior to enrollment and no additional treatment during the study; 2) non-melanoma skin cancer or malignant freckle-like sputum with adequate treatment and no evidence of disease recurrence; 3) adequately treated and In situ carcinoma without evidence of disease recurrence;
* Female patients who are pregnant or breastfeeding
* According to the investigator's judgment, there are serious concomitant diseases that endanger the safety of the patient or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | From first treatment，each 42 or 63 days until PD or death(up to 24 months)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 42 or 63 days until intolerant the toxicity or PD (up to 24 months) ]
Disease Control Rate (DCR) | each 42 or 63 days until intolerant the toxicity or PD (up to 24 months) ]
Duration of Response(DOR) | each 42 or 63 days until intolerant the toxicity or PD (up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: LUO SUXIA, Study Chair — Henan Cancer Hospital
Locations (6):
- China (6):
  - ANYANG Cancer Hospital, Anyang, Henan
  - First Affiliated Hospital of Henan University of Science and Technolog, Luoyan, Henan
  - Henan cancer hospital, Zhengzhou, Henan
  - Qilu Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Central Hospital, Linyi, Shandong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li N, Wu T, Hong YG, Guo YZ, Cheng YF, Ma YJ, Bie LY, Cui DH, Gao XH, Tan BX, Li BS, Luo SX, Wang JS. A multi-center, single-arm, phase II study of anlotinib plus paclitaxel and cisplatin as the first-line therapy of recurrent/advanced esophageal squamous cell carcinoma. BMC Med. 2022 Dec 8;20(1):472. doi: 10.1186/s12916-022-02649-x. PMID 36482345